CLINICAL TRIAL: NCT06396481
Title: Clinical Study of Allogeneic Vγ9Vδ2 T Cells in the Treatment of Brain Malignant Glioma
Acronym: CSAγδTBMG
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX-A-2022006-1
Record Dates: First submitted 2024-03-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: GBM; DIPG Brain Tumor; Medulloblastoma
Keywords: malignant glioma; Vγ9Vδ2 T
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Medulloblastoma; Glioma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- To evaluate the safety and feasibility of allogeneic Vγ9Vδ2 T cell therapy. (Experimental): The trial consisted of two phases: dose climbing phase and extension phase. At least 15 patients with malignant brain glioma (WHO Grade IV) were enrolled in the climbing phase. According to the 3+3 design, the amount of cells suitable for implantable Ommaya capsules for cell transfusion was increased according to the dose of 1x107, 3x107, 1x108 and 3x108 per dose, so as to observe its tolerability and safety. In the expansion phase, 10 patients with malignant brain glioma (WHO Grade IV) were enrolled, and dose expansion therapy was performed according to the optimal dose obtained in the climbing phase to observe its tolerability and safety. One course of treatment every 4 weeks, a total of 3 courses. Vγ9Vδ2 T cells were injected into the ventricle or ventricle once a week for the first three weeks and observed at the fourth week. In some patients, radiotherapy or other chemotherapy drugs (such as temozolomide) may be combined at week 4.
  Interventions: Biological: Vγ9Vδ2 T cell
- To evaluate the therapeutic effect of allogeneic Vγ9Vδ2 T cells on brain malignant glioma (Experimental): The trial consisted of two phases: dose climbing phase and extension phase. At least 15 patients with malignant brain glioma (WHO Grade IV) were enrolled in the climbing phase. According to the 3+3 design, the amount of cells suitable for implantable Ommaya capsules for cell transfusion was increased according to the dose of 1x107, 3x107, 1x108 and 3x108 per dose, so as to observe its tolerability and safety. In the expansion phase, 10 patients with malignant brain glioma (WHO Grade IV) were enrolled, and dose expansion therapy was performed according to the optimal dose obtained in the climbing phase to observe its tolerability and safety. One course of treatment every 4 weeks, a total of 3 courses. Vγ9Vδ2 T cells were injected into the ventricle or ventricle once a week for the first three weeks and observed at the fourth week. In some patients, radiotherapy or other chemotherapy drugs (such as temozolomide) may be combined at week 4.
  Interventions: Biological: Vγ9Vδ2 T cell
- To investigate the expansion, infiltration and persistence of Vγ9Vδ2 T cells after reinfusion. (Experimental): The trial consisted of two phases: dose climbing phase and extension phase. At least 15 patients with malignant brain glioma (WHO Grade IV) were enrolled in the climbing phase. According to the 3+3 design, the amount of cells suitable for implantable Ommaya capsules for cell transfusion was increased according to the dose of 1x107, 3x107, 1x108 and 3x108 per dose, so as to observe its tolerability and safety. In the expansion phase, 10 patients with malignant brain glioma (WHO Grade IV) were enrolled, and dose expansion therapy was performed according to the optimal dose obtained in the climbing phase to observe its tolerability and safety. One course of treatment every 4 weeks, a total of 3 courses. Vγ9Vδ2 T cells were injected into the ventricle or ventricle once a week for the first three weeks and observed at the fourth week. In some patients, radiotherapy or other chemotherapy drugs (such as temozolomide) may be combined at week 4.
  Interventions: Biological: Vγ9Vδ2 T cell

INTERVENTIONS:
Biological: Vγ9Vδ2 T cell — The trial consisted of two phases: dose climbing phase and extension phase. At least 15 patients with malignant brain glioma (WHO Grade IV) were enrolled in the climbing phase. According to the 3+3 design, the amount of cells suitable for implantable Ommaya capsules for cell transfusion was increased according to the dose of 1x107, 3x107, 1x108 and 3x108 per dose, so as to observe its tolerability and safety. In the expansion phase, 10 patients with malignant brain glioma (WHO Grade IV) were enrolled, and dose expansion therapy was performed according to the optimal dose obtained in the climbing phase to observe its tolerability and safety. One course of treatment every 4 weeks, a total of 3 courses. Vγ9Vδ2 T cells were injected into the ventricle or ventricle once a week for the first three weeks and observed at the fourth week. In some patients, radiotherapy or other chemotherapy drugs (such as temozolomide) may be combined at week 4.

SUMMARY:
Primary brain malignant tumor has become the first lethal tumor in children and young adults, and the treatment is limited, and the prognosis of patients is poor. According to the classification of the World Health Organization, glioblastoma is divided into grade II, III and IV gliomas; The higher the degree of malignancy, the worse the clinical outcome. Among them, the most malignant, most lethal, and most common types of tumors include supratentorial glioblastoma, diffuse endopontine glioma (DIPG), medulloblastoma, and ependymoma. Its high malignancy is mainly manifested in three aspects: extremely rapid growth and obvious invasion; The operation is not easy to remove all; The tumor has a tendency of recurrence and disseminated implantation. It can occur with children and adults of all ages. At present, surgery combined with chemoradiotherapy is the main treatment, but the therapeutic effect is not good. Studies have shown that glioblastoma, as the most common primary brain malignant tumor in adults, after standard surgery, radiotherapy and chemotherapy, the median survival time is less than 15 months, and the overall five-year survival rate is only 5.4%. Even after receiving new and expensive Tumor-treating fields, the median survival time is less than 21 months. The median survival time of DIPG patients is generally less than 1 year, and the 5-year survival rate is less than 5%. The average 5-year survival rate of medulloblastoma and anaplastic ependymoma is 40%~60%. Innovative treatments are urgently needed. Immunotherapy based on Vγ9Vδ2 T cells has become a promising research direction in recent years. Its unique phosphine antigen recognition does not depend on major histocompatibility complex (MHC), easy to allograft and other advantages. Making it one of the most promising cell therapies. Brain glioma has abnormal cholesterol metabolism and phosphine antigen accumulation, which is easily sensed by Vγ9Vδ2 T cells. Therefore, the clinical exploration of Vγ9Vδ2 T cells for glioma is of great significance to both the scientific and clinical communities.

DETAILED DESCRIPTION:
Research purpose

1. Main purpose:

   To evaluate the safety and feasibility of allogeneic Vγ9Vδ2 T cell therapy.
2. Secondary Purpose:

   To evaluate the therapeutic effect of allogeneic Vγ9Vδ2 T cells on brain malignant glioma (WHO IV).
3. Explore goals:

To investigate the expansion, infiltration and persistence of Vγ9Vδ2 T cells after reinfusion. To investigate the immunological dynamics of Vγ9Vδ2 T cells after reinfusion. To explore biomarkers that might predict the clinical efficacy of Vγ9Vδ2 T cell therapy.

Research design types, principles and test steps

1. Research design This is an exploratory clinical trial. It is planned to enroll 50 patients with malignant glioma (WHO Grade IV) in the Department of Neurosurgery of Beijing Tiantan Hospital to conduct a single-center, single-arm open phase I clinical trial. To evaluate the safety, feasibility, and efficacy of allogeneic Vγ9Vδ2 T cell infusion regimen in the treatment of malignant brain gliomas (WHO Grade IV).

   The trial consisted of two phases: dose climbing phase and extension phase. At least 15 patients with malignant brain glioma (WHO Grade IV) were enrolled in the climbing phase. According to the 3+3 design, the cell transfusion volume was successively increased according to the doses of 1x107, 3x107, 1x108 and 3x108 per dose to observe its tolerability and safety. In the expansion phase, 10 patients with malignant brain glioma (WHO Grade IV) were enrolled, and dose expansion therapy was performed according to the optimal dose obtained in the climbing phase to observe its tolerability and safety. One course of treatment every 4 weeks, a total of 3 courses. At the same time, patients who failed to complete at least one course of precision treatment for any reason after enrollment were included in the internal control group, and patients who met the admission criteria of this study but did not participate in this study were included in the external control group, with a total of 25 cases.
2. Sample size and research plan After signing the informed consent form (ICF), subjects will complete the screening period assessment according to the trial plan process sheet. Patients can be combined with the chemotherapy drug temozolomide according to the specific condition.

Recruit 20 healthy donors to provide peripheral blood. After the donors sign the informed consent, they will complete the evaluation and collection of peripheral blood according to the procedure table of the trial plan.

After screening qualified donors, it is necessary to arrange monopexing as soon as possible. The full name of mononuclear cell collection is peripheral blood mononuclear cell collection. In this study, blood cell separation will be used for mononuclear cell collection.

Monofrequency: ECG monitoring was performed before and during monofrequency, and was recorded once an hour from the beginning until the end of monofrequency. The collection time must record the circulation amount, collection volume, and collection time in a timely manner. Information on the preparation of single samples and Vγ9Vδ2 T cells was collected and recorded. If the donor does not consent to the continued use of its Vγ9Vδ2 T cells in this study, the study will be destroyed in accordance with the standard procedures prescribed by national law.

At least 15 patients with malignant brain glioma (WHO Grade IV) were initially planned to be enrolled using a staggered dosing strategy. Subject 1 and 2, and subject 2 and 3 must be monitored at least 2 weeks apart. The number of allogeneic Vγ9Vδ2 T cells was increased at each dose of 1×107, 3×107, 1×108, and 3x108 to observe their tolerance and safety. Short-term safety evaluation was performed 2-3 days after each course of cell infusion. After the treatment, according to the number of successfully prepared allogeneic Vγ9Vδ2 T cells, the study doctor can choose to continue to give cell transfusion for multiple courses according to the clinical condition of the subjects.

Further enrollment of 10 patients with malignant brain glioma (WHO Grade IV) is planned for dose-extension therapy at the optimal dose obtained above to observe tolerability and safety. One course of treatment every 4 weeks, a total of 3 courses. Short-term safety evaluation was performed 2-3 days after each course of cell infusion. After the end of 3 courses, the number of successfully prepared Vγ9Vδ2 T cells can also be selected by the research doctor according to the clinical condition of the subjects to continue to give cell transfusion for multiple courses. Patients who failed to complete at least one course of precision treatment for any reason after enrollment were included in the internal control group, and patients who met the admission criteria of this study but did not participate in this study were included in the external control group, with a total of 25 cases.

Follow-up was performed at 30 days, 2 months, 3 months, 6 months, 9 months, and 12 months after the first cell reinfusion, or early withdrawal from the study, and efficacy was assessed at each follow-up.

The end of the trial was defined as withdrawal of informed consent by the last subject, termination of treatment or withdrawal from the trial, loss of follow-up or death, completion of 1 year of follow-up, or early termination of the study, whichever occurred first.

The trial may be terminated prematurely at any time for any reason attributable to the Sponsor. If necessary, the subject should have an end-of-treatment visit as soon as possible.

4. Research methods Vγ9Vδ2 T cell therapy program

This is an exploratory clinical trial. It is planned to enroll 50 patients with malignant glioma (WHO Grade IV) in the Department of Neurosurgery of Beijing Tiantan Hospital to conduct a single-center, single-arm open phase I clinical trial. To evaluate the safety, feasibility, and efficacy of allogeneic Vγ9Vδ2 T cell infusion regimen in the treatment of malignant brain gliomas (WHO Grade IV).

The trial consisted of two phases: dose climbing phase and extension phase. At least 15 patients with malignant brain glioma (WHO Grade IV) were enrolled in the climbing phase. According to the 3+3 design, the amount of cells suitable for implantable Ommaya capsules for cell transfusion was increased according to the dose of 1x107, 3x107, 1x108 and 3x108 per dose, so as to observe its tolerability and safety. In the expansion phase, 10 patients with malignant brain glioma (WHO Grade IV) were enrolled, and dose expansion therapy was performed according to the optimal dose obtained in the climbing phase to observe its tolerability and safety. One course of treatment every 4 weeks, a total of 3 courses. Vγ9Vδ2 T cells were injected into the ventricle or ventricle once a week for the first three weeks and observed at the fourth week. In some patients, radiotherapy or other chemotherapy drugs (such as temozolomide) may be combined at week 4.

The study was a single-arm, single-center intervention Phase I clinical study. The overall study was carried out in two steps:

1. Uphill phase: At least 15 patients with malignant glioma (WHO Grade IV) were initially planned to be enrolled. According to the 3+3 design, the amount of cell transfusion was increased successively according to the doses of 1x107, 3x107, 1x108 and 3x108 per dose to observe the tolerance and safety of the cells.
2. Expansion stage: 10 patients with malignant brain glioma (WHO Grade IV) are planned to be enrolled for dose expansion therapy according to the optimal dose obtained in the climbing stage, so as to observe its tolerability and safety. One course of treatment every 4 weeks, a total of 3 courses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed malignant brain glioma in an important structural area (WHO Grade IV);
* Patients with poor postoperative effect or ineffective guidelines for conventional treatment
* Age ≥4 years old, male or female;
* KPS score ≥70;
* Normal bone marrow reserve function and normal liver and kidney function (as evidenced by the following laboratory tests prior to initial Vγ9Vδ2 T cell therapy) :
* Neutrophil absolute value ≥ 1,500/mm3;
* hemoglobin 10g/dL;
* Platelet count > 100,000/mm3;
* Glutamic pyruvic transaminase/Glutamic oxalacetic transaminase < 2.5 x ULN;
* Serum creatinine 1.5×ULN;
* Total bilirubin levels < 1.5 x ULN.
* No obvious genetic diseases;
* Normal cardiac function, cardiac ejection index > 55%;
* Suitable for implantation of Ommaya capsule in ventricle or cavity;
* No bleeding and coagulation disorders;
* Women of reproductive age (15-49 years) must undergo a negative pregnancy test within 7 days before starting treatment and use contraception during the clinical trial period and within 3 months after the last cell transfusion;
* Sign the informed consent form.

Exclusion Criteria:

* Pregnant and lactating women;
* Organ failure;
* Heart: Grade III and grade IV;
* Liver: Level C of the Child-Turcotte liver function scale;
* Kidney: renal failure and uremia stage;
* Lungs: Symptoms of severe respiratory failure;
* Brain: A person with a disorder of consciousness.
* Patients with a history of organ transplantation;
* Uncontrollable infectious disease or other serious illness, including but not limited to infection (such as HIV positive), congestive heart failure, unstable angina pectoris, arrhythmia, psychosis, or restrictive social environment or what the attending physician considers to be an unpredictable risk;
* Patients with systemic autoimmune disease or immunodeficiency;
* Patients with allergic constitution;
* Use of systemic steroid drugs;
* Have a chronic disease that requires the use of immune agents or hormone therapy;
* Prior treatment with any other immune cell;
* Have participated in other clinical trials within the past 30 days;
* The researchers believe that other reasons are not suitable for clinical trials

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | up to 12 months
  The study will collect all adverse events that occurred after participants initiated leukocyte monopexy to Vγ9Vδ2 T cell therapy for a specified period of time or until disease progression. Safety assessment tests include: blood oxygen saturation should not be lower than 80mmHg; The ECG results of heart rate and ECG should be normal sinus rhythm. Blood biochemical examination of white blood cells should be maintained at 4000-10000/μL level; IL6 should be less than 200pg/mL. Safety assessment was performed according to the study protocol one day before each infusion of Vγ9Vδ2 T cells and one week after each infusion. Safety assessment tests include: blood oxygen saturation should not be lower than 80mmHg; The ECG results of heart rate, PR interval, RR interval, QRS, QT interval, QTcF and ECG should be normal sinus rhythm. Blood biochemical examination of white blood cells should be maintained at 4000-10000/μL level; IL6 should be less than 200pg/mL.

SECONDARY OUTCOMES:
curative effect appraising | up to 12 months
  Primary endpoints typically included MRI measurements of enhanced lesions in the lumen before and each week after reinfusion using RANO criteria: complete response (disappearance of enhanced lesions), partial response (reduction > 30%), disease stabilization (reduction <30% or increase < 20%), or disease progression (lesions > 20% or emergence of new lesions).
  Survival analysis: Overall survival (OS), which measures the time from the start of treatment to death from any cause, is measured in months, compared to historical controls, and has an effect of 14 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Sun, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No